CLINICAL TRIAL: NCT07397130
Title: Inspiratory Muscle Pressure and Diaphragmatic Strength in Women With Long COVID-19: A Pressure Biofeedback-Guided Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSUP Persahabatan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0171/KEPK-RSUPP/07/2024
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Long COVID-19 Syndrome; Post COVID Syndrome Long Covid; Post COVID-19 Syndrome
Keywords: Post Covid; Diaphragmatic Strength; Inspiratory Pressure; Pressure Biofeedback Exercise; Pulmonary Rehabilitation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Control Group (Standard rehabilitation) and Intervention Group (Pressure biofeedback exercise)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group receive indirect diaphragmatic muscle training using pressure biofeedback as part of post-COVID-19 respiratory rehabilitation. The training is performed using a pressure biofeedback unit placed at the lumbosacral region to provide real-time feedback during diaphragmatic breathing exercises. Participants are instructed to perform controlled diaphragmatic breathing aimed at increasing abdominal expansion while minimizing chest wall movement. The exercise program is conducted according to a structured protocol over the intervention period to improve diaphragmatic muscle activation, increase inspiratory muscle strength, and enhance maximal inspiratory pressure.
  Interventions: Device: Pressure Biofeedback Unit
- Control Group (No Intervention): Participants receive standard post-COVID-19 care without indirect diaphragmatic muscle training using pressure biofeedback. No structured pressure biofeedback-guided diaphragmatic training is provided during the study period.

INTERVENTIONS:
Device: Pressure Biofeedback Unit — Diaphragmatic muscle training using a pressure biofeedback unit is provided as part of post-COVID-19 respiratory rehabilitation. The pressure biofeedback unit is placed at the lumbosacral region to provide real-time feedback during diaphragmatic breathing exercises. Participants are instructed to perform controlled diaphragmatic breathing aimed at enhancing diaphragmatic activation and increasing inspiratory muscle strength.
  Arms: Intervention Group

SUMMARY:
COVID-19 is an infectious disease that can cause long-term health problems even after the acute infection has resolved. Many people who have recovered from COVID-19 continue to experience breathing difficulties, fatigue, and reduced physical capacity. These ongoing problems are often related to decreased lung function and weakness of the breathing muscles, especially the diaphragm, which plays a major role in breathing.

In women after COVID-19, respiratory muscle weakness may result from inflammation during infection, prolonged bed rest, and increased effort required to breathe. This can lead to reduced inspiratory strength, shortness of breath, and limitations in daily activities. Respiratory rehabilitation is therefore important to help restore breathing muscle strength and improve overall respiratory function.

One rehabilitation approach is indirect diaphragmatic muscle training using pressure biofeedback. This method provides visual or tactile feedback during breathing exercises to help patients activate and strengthen the diaphragm more effectively. Pressure biofeedback has been used as part of post-COVID-19 rehabilitation in Indonesia, but its effectiveness in improving inspiratory strength and diaphragmatic function, particularly in women after COVID-19, has not been fully evaluated.

The purpose of this study is to examine the relationship between improvements in maximal inspiratory pressure and improvements in diaphragmatic strength in women recovering from COVID-19 who perform indirect diaphragmatic muscle training using pressure biofeedback. The study hypothesizes that indirect diaphragmatic training guided by pressure biofeedback can improve diaphragmatic strength and increase maximal inspiratory pressure in women after COVID-19.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19), caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), has resulted in a growing population of individuals experiencing persistent symptoms after the acute phase of infection. Post-COVID-19 conditions frequently involve respiratory impairment, characterized by reduced lung capacity, decreased maximal inspiratory pressure, and weakness of the respiratory muscles, particularly the diaphragm. These impairments are attributed to systemic inflammation, cytokine storm, prolonged immobilization, increased respiratory workload, and neuromuscular involvement during and after COVID-19 infection.

The diaphragm is the primary inspiratory muscle and plays a critical role in maintaining adequate ventilation. Diaphragmatic dysfunction following COVID-19 may manifest as reduced diaphragmatic excursion, decreased muscle thickness, and diminished inspiratory pressure generation. Maximal inspiratory pressure (MIP) is a widely used, non-invasive parameter for assessing inspiratory muscle strength and reflects the functional capacity of the diaphragm and accessory inspiratory muscles. Reduced MIP values indicate inspiratory muscle weakness and are associated with impaired respiratory function and reduced physical capacity.

Women after COVID-19, particularly in the postpartum period, represent a vulnerable population for respiratory muscle weakness. Physiological changes related to pregnancy and childbirth, combined with the effects of COVID-19 infection, may exacerbate diaphragmatic weakness and impair respiratory mechanics. Despite the clinical relevance of this condition, data regarding targeted respiratory rehabilitation interventions in this population remain limited.

Respiratory rehabilitation has been shown to improve respiratory muscle strength, reduce dyspnea, and enhance quality of life in post-COVID-19 patients. One rehabilitation approach is indirect diaphragmatic muscle training using pressure biofeedback. This technique utilizes a pressure-sensing device placed at the lumbosacral region to provide real-time feedback during diaphragmatic breathing exercises. The feedback allows patients to optimize diaphragmatic activation while minimizing excessive chest wall movement, thereby promoting effective and controlled diaphragmatic contraction.

Indirect diaphragmatic training with pressure biofeedback is designed to strengthen the diaphragm by encouraging abdominal expansion during inspiration. Repeated training sessions aim to increase diaphragmatic endurance and strength, leading to improvements in maximal inspiratory pressure and overall respiratory function. This method has been used in respiratory rehabilitation settings in Indonesia; however, its specific effectiveness in improving diaphragmatic strength and inspiratory pressure in women after COVID-19 has not been adequately studied.

This study employs a randomized, single-blind clinical trial design to evaluate the relationship between changes in maximal inspiratory pressure and changes in diaphragmatic strength following indirect diaphragmatic muscle training using pressure biofeedback. Participants are allocated to either a control group or an intervention group. The intervention group receives structured indirect diaphragmatic training with pressure biofeedback over a defined training period, while both groups undergo standardized assessments of inspiratory pressure and diaphragmatic muscle function at predetermined time points.

Diaphragmatic strength is assessed using ultrasonographic evaluation of diaphragmatic movement and thickness, while maximal inspiratory pressure is measured using a pressure manometer. These measurements allow for objective evaluation of respiratory muscle function and enable analysis of the correlation between inspiratory pressure improvement and diaphragmatic muscle strengthening following the intervention.

The primary scientific focus of this study is to determine whether improvements in maximal inspiratory pressure are correlated with improvements in diaphragmatic strength following indirect diaphragmatic muscle training guided by pressure biofeedback. By examining this relationship, the study aims to provide evidence supporting the role of pressure biofeedback-guided diaphragmatic training as a respiratory rehabilitation modality for women recovering from COVID-19.

The findings of this study are expected to contribute to the development of evidence-based respiratory rehabilitation strategies for post-COVID-19 conditions, particularly in women, and to support the integration of pressure biofeedback techniques into comprehensive post-COVID-19 rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Female patients treated at Persahabatan Hospital.
* History of COVID-19 infection.
* Attending the Pulmonology Clinic and/or the Medical Rehabilitation Clinic at Persahabatan Hospital.
* Willing to participate in indirect diaphragmatic training using pressure biofeedback for four consecutive weeks.
* Willing to participate as research subjects.

Exclusion Criteria:

* Female patients not treated at Persahabatan Hospital
* No history of COVID-19 infection
* Not participating in indirect diaphragmatic training using pressure biofeedback for four consecutive weeks
* Presence of other pulmonary disease such as tuberculosis, chronic obstructive pulmonary disease, or asthma

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic Muscle Strength | Baseline and after completion of the intervention period (at 4 weeks)
  Diaphragmatic muscle strength is assessed using ultrasonographic evaluation of diaphragmatic movement and thickness during respiration to determine diaphragmatic function.
Maximal Inspiratory Pressure (MIP) | Baseline and after completion of the intervention period (at 4 weeks)
  Maximal inspiratory pressure is measured to assess inspiratory muscle strength. MIP is evaluated using a pressure manometer during a maximal inspiratory effort and reflects the functional strength of the diaphragm and other inspiratory muscles.
Maximal Expiratory Pressure (MEP) | Baseline and after completion of the intervention period (at 4 weeks)
  Maximal expiratory pressure is measured to assess expiratory muscle strength. MEP is evaluated using a pressure manometer during a maximal expiratory effort and reflects the strength of the abdominal and expiratory respiratory muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Umum Pusat Persahabatan, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Study Outcome
Supporting Information: Study Protocol
Time Frame: 4 weeks
Access Criteria: by request to my email: sitichandraw@gmail.com